CLINICAL TRIAL: NCT05311033
Title: Evaluation of a Tranexamoc Acid Treatment on Post-inflammatory Pigmentation Induced in the Suction Blister Model - Study HPPI
Brief Title: Evaluation of a Tranexamoc Acid Treatment on Post-inflammatory Pigmentation in the Suction Blister Model
Acronym: TRANEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-PP-07
Record Dates: First submitted 2022-03-07; First posted 2022-04-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Skin Pigmentation
MeSH Terms: conditions — Pigmentation Disorders | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Samples Without DNA (Experimental): Healthy males aged 20-40 years with at risk of post-inflammatory hyperpigmentation: phototype IV or V according to the Fitzpatrick scale (1) and having a colorimetric individual typology angle (ITA°) between -20° and 28° and/or having already had post-inflammatory pigmentation or hyperpigmentation (e.g. acne scars, melasma)
  Interventions: Other: Exacyl

INTERVENTIONS:
Other: Exacyl — Healthy males with at risk of post-inflammatory hyperpigmentation have a skin samples for evaluate the activity of tranexamic acid.

SUMMARY:
Post-inflammatory hyperpigmentation (PIH) is a common sequela of inflammatory dermatoses. PIH results from the overproduction of melanin or irregular pigment dispersion after skin inflammation. The investigators have developed, validated and published an in vivo model of PIH based on an initial lesion involving suction blisters. In this study, they have demonstrated that the suction blisters model is able to reproduce an epidermal lesion and inflammatory state that, in melanin competent subjects, leads to consistent hyperpigmentation during real sunlight exposure without the need for additional artificial exposure to intense UV light.

An increase in vascularisation is demonstrated by histology in early forms of PIH. The investigators have also shown this increase in vascularisation in their PIH model. Furthermore, the transcriptomic study in this model shows that UVA and visible light directly stimulate endothelial cells and increase angiogenesis but act essentially indirectly through the production by fibroblasts of uPA (urokinase-type plasminogen activator), a key factor in the modulation of extracellular matrices, inflammatory processes and angiogenesis.

UPA is a serine protease that converts plasminogen to plasmin which promotes angiogenesis. Tranexamic acid (TA) is an antifibrinolytic that reversibly binds to plasminogen, preventing its conversion to plasmin and subsequent fibrin degradation.

The aim of the study will be to evaluate the efficacy of tranexamic acid in preventing post-inflammatory hyperpigmentation induced in the suction blisters model in at-risk subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who has signed and dated an information and informed consent form before any study-related procedure is initiated,
2. A healthy male subject between the ages of 20 and 40 years
3. Subject at risk of HPPI: phototype IV or V according to the Fitzpatrick scale (1) and having a colorimetric individual typology angle (ITA°) between -20°/ and 28° and/or having previous post-inflammatory gold pigmentation or hyperpigmentation (e.g. acne scars, melasma)
4. Subjects willing to undergo skin biopsies and who do not have any contraindications related to biopsy procedures such as allergy to local anaesthetics or local antiseptics (Chlorhexidine), coagulation problems, having an anticoagulant treatment or a history of wound healing problems or vasovagal hypotension or syncope.
5. Subject willing to follow the study restrictions and willing to complete the study,
6. Subject covered by a Social Security scheme in accordance with the Public Health Code (Article L1121-11)

Exclusion Criteria:

1. Subjects with contraindications to tranexamic acid :

   * Subjects allergic to tranexamic acid or to any of the other components contained in Exacyl,
   * Subject suffering from arterial or venous thrombosis,
   * Subjects with a history of thromboembolic disease or with an increased incidence of thromboembolic events in their family history (patients at high risk of thrombophilia)
   * Subjects with consumer coagulopathy,
   * Subjects with kidney problems,
   * Subjects with a history of seizures
   * Subjects allergic to wheat as Exacyl contains wheat starch
   * Subject with fructose intolerance, glucose-galactose malabsorption syndrome or sucrase/isomaltase deficiency
2. Subjects with active systemic or skin disease that could in any way interact with the interpretation of the study results (e.g. atopic dermatitis or psoriasis),
3. Subjects who are planning to be exposed to intense sunlight during the study or who have been exposed within 6 weeks prior to the screening visit,
4. Subject having used any anti-inflammatory product (steroidal and non-steroidal anti-inflammatory drugs) for more than 5 consecutive days in the month prior to inclusion or having planned to use these drugs during the study,
5. Subjects taking treatments known to be active on skin healing,
6. Subjects with a significant history of alcohol or drug abuse or with a psychotic state,
7. Subject with a history of keloids or hypertrophic scars,
8. Subject with a positive hepatitis B, hepatitis C or HIV status at the screening visit,
9. Subject with a history of serious illness (based on the subject's history and/or the results of the screening physical examination) that, in the opinion of the Investigator, would place the subject at risk by participating in the study or would significantly interfere with the evaluation of the study outcome (e.g. cancer, immunity disorder),
10. Subjects who are hospitalised in a medical or social institution for any reason other than biomedical research or who have lost their liberty by administrative or legal decision or who are under guardianship,
11. Subject unable to communicate or cooperate with the Investigator due to mental impairment, language problems or impaired brain function,
12. Subject who has received treatment with a non-marketed substance in the 4 weeks prior to inclusion or longer, if the substance family requires a longer wash-out period,
13. Subject who has received (or will receive) more than 4500 euros in compensation for participation in clinical studies during the 12 months preceding the study.
14. Subjects protected by law

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline post-inflammatory hyperpigmentation induced in the suction blister model Systolic Blood Pressure at 6 months | at Day 1 (baseline) and 72 days
  To evaluate the activity of tranexamic acid on the prevention of post-inflammatory hyperpigmentation induced in the suction blister model in subjects at risk

SECONDARY OUTCOMES:
The number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | at Day 29 and Day 64
  To evaluate the tolerance and possible adverse effects during 5 weeks of tranexamic acid treatment on post-inflammatory hyperpigmentation induced in the suction blister model

CONTACTS AND LOCATIONS:
Overall Officials: passeron thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No